CLINICAL TRIAL: NCT01974011
Title: Comparison of Dorsal Penile Nerve Block (DPNB According to Dalens' Technique) to Dorsale Penile Nerve Block With Ventromedial Infiltration
Brief Title: DPNB vs. Modified DPNB With Ventromedial Infiltration (DPNB According to Dalens' Technique)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care - Medicine CVK/CCM, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPNB vs. Modified DPNB
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Circumcision, Meatotomy or Distal Coronary Correction of Hypospadia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dorsal penile nerve block according to Dalens' technique (Experimental): Two injections at the dorsum penis according to Dalens' technique.
  Interventions: Procedure: Performing dorsal penile nerve block (DPNB)
- DPNB with additional infiltration of the ventromedial penis (Active Comparator): Modified procedure:
  Two injections at the dorsum penis according to Dalens' technique plus on subcutaneous injection in the ventral midline of the penis at the transition between the penis and the scrotum.
  Interventions: Procedure: Performing dorsal penile nerve block (DPNB)

INTERVENTIONS:
Procedure: Performing dorsal penile nerve block (DPNB)

SUMMARY:
Dorsal penile nerve block (DPNB) is a regional nerve block probably most often performed throughout the world. There are several different methods described in the literature. When compared to penile ring wall infiltration or caudal block, the Dorsal penile nerve block (DPNB) is more likely associated with the risk of failure of the block quality. The aim of this study is to compare the quality of the standard method of Dorsal penile nerve block (DPNB)(Dalens' technique) with that of a modified procedure (Dorsal penile nerve block (DPNB)with additional infiltration of the ventromedial penis at the transition between the penis and the scrotum.

DETAILED DESCRIPTION:
Male circumcision is the most often performed operation in male children throughout the world. In the western world it is not accepted to perform this procedure without adequate analgesic support. Hence the dorsal penile nerve block (DPNB), first described in the 70ies of the 20th century, is one of the most frequently performed regional anesthetic procedures in both children and adults. There are several methods described in the literature, of which the one described by Dalens et al in 1989 nowadays is the most often quoted and most frequently performed method. The reported rate of insufficient analgesia by DPNB is higher than caudal block or penile ring wall infiltration. It is known from neuroanatomic studies, that the penis is innervated mostly, but not only by the dorsal penile nerve, a final branch of the pudendal nerve. A varying amount of the ventral penile skin, especially of the preputium and the frenulum, is innervated by fine end branches of the perineal nerve, which otherwise gives sensoric innervation to the scrotum and motor innervation to the bulbospongiosus muscle. An injection of local anesthetic underneath Buck's fascia is unable to reach the perineal nerve, which may be the explanation for these failures.

In this study we compare two different techniques of performing the dorsal penile nerve block (DPNB): the technique according to Dalens, and a modification, where a small amount of the local anesthetic for the dorsal penile nerve block (DPNB) is withheld, and then injected subcutaneously at the ventral transition between the penis and the scrotum in the midline. The latter injection at the site of perineal innervation is a relic of the penile ring wall infiltration, which surely blocks all skin fibres of both the dorsal penile nerve and the perineal nerve.

All patients included randomly receive either two injections at the dorsum penis according to Dalens' technique, or two injections at the dorsum penis according to Dalens' technique plus on subcutaneous injection in the ventral midline of the penis at the transition between the penis and the scrotum. The amount of local anesthetic (bupivacaine 0,75%, 0,2 ml/kg of body weight) and dosing of narcotics (Sevoflurane 2,2 Vol% end-expiratory gas in an oxygen-air mixture) is the same in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Male infant
* Aged 1-17 years
* Elective surgery for circumcision, meatotomy or distal coronary correction of hypospadia

Exclusion Criteria:

* Allergy to local anaesthetics
* Sepsis
* Congenital or acquired bleeding disorders
* Neurological disease
* Significant damage of central nervous system
* Other malformation of urethra

Ages: 1 Year to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2016-01-05 (Actual); Study Completion 2016-01-06 (Actual)

PRIMARY OUTCOMES:
Need for opioid analgesics | On the day of surgery

SECONDARY OUTCOMES:
Need for analgesics | Perioperatively up to the seventh postoperative day
Pain | perioperatively up to the seventh postoperative day
  Incidence and severity of pain
Hospital length of stay | Up to hospital discharge, an exspected average of one day
Length of stay within post-anesthesia recovery unit | Up to post-anesthesia recovery unit discharge, an exspected average of six hours
Postoperative complications and infections | Perioperatively up to the seventh postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Berlin, Germany

REFERENCES:
- [Background] Dalens B, Vanneuville G, Dechelotte P. Penile block via the subpubic space in 100 children. Anesth Analg. 1989 Jul;69(1):41-5. PMID 2742166
- [Background] Long RM, McCartan D, Cullen I, Harmon D, Flood HD. A preliminary study of the sensory distribution of the penile dorsal and ventral nerves: implications for effective penile block for circumcision. BJU Int. 2010 Jun;105(11):1576-8. doi: 10.1111/j.1464-410X.2009.09044.x. Epub 2009 Nov 4. PMID 19889061
- [Background] Serour F, Mori J, Barr J. Optimal regional anesthesia for circumcision. Anesth Analg. 1994 Jul;79(1):129-31. doi: 10.1213/00000539-199407000-00024. PMID 8010422
- [Background] Stav A, Gur L, Gorelik U, Ovadia L, Isaakovich B, Sternberg A. Modification of the penile block. World J Urol. 1995;13(4):251-3. doi: 10.1007/BF00182973. PMID 8528302
- [Background] Szmuk P, Ezri T, Ben Hur H, Caspi B, Priscu L, Priscu V. Regional anaesthesia for circumcision in adults: a comparative study. Can J Anaesth. 1994 Dec;41(12):1181-4. doi: 10.1007/BF03020658. PMID 7867113
- [Background] Weksler N, Atias I, Klein M, Rosenztsveig V, Ovadia L, Gurman GM. Is penile block better than caudal epidural block for postcircumcision analgesia? J Anesth. 2005;19(1):36-9. doi: 10.1007/s00540-004-0287-8. PMID 15674514
- [Background] Yucel S, Baskin LS. Neuroanatomy of the male urethra and perineum. BJU Int. 2003 Oct;92(6):624-30. doi: 10.1046/j.1464-410x.2003.04435.x. PMID 14511049